CLINICAL TRIAL: NCT04925154
Title: PATHOS Tradeoffs in Patient Decision Making About Rectal Cancer Treatment: Benefits Compared to Quality Of Life.
Brief Title: Tradeoffs in Patient Decision Making About Rectal Cancer Treatment: Benefits Compared to Quality Of Life.
Acronym: Pathos
Status: Recruiting | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Te Vuong, Radiation-oncologist, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: 2021-2517
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Patient Preference
Keywords: Colorectal cancer; Treatment preferences
MeSH Terms: conditions — Patient Preference; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients: Recruitment for this group will take place at either the radiation-oncology department or at the colorectal surgery department, at the time of consultation or at the time of diagnosis, before the treatment setting. Once clinical staging is available, the surgeon and/or radiation-oncologist and/or research assistant should identify eligible patients. Patients that comply with selection criteria (inclusion/exclusion) will be approached by a research team member. For those patients interested in participating, the e-link to the consent form for this group will be sent by email. Once a patient decides to sign the consent form, the link for the questionnaire Q1 will be sent by email.
  Interventions: Behavioral: The only intervention will be the information brochure that will be given after the first questionnaire.
- Group B: Physicians: Health professionals will be approached by the research team. The study aim will be explained, and participants that agree to participate will be provided an e-link to consent for this group. Once the health care participant decides to sign the consent form, the link for the questionnaire Q1 will be sent by email.
  Interventions: Behavioral: The only intervention will be the information brochure that will be given after the first questionnaire.

INTERVENTIONS:
Behavioral: The only intervention will be the information brochure that will be given after the first questionnaire. — The information brochure will be given to both groups at the same time at 2-3 weeks after the first consultation (patients group) or after answering the first questionnaire (physicians group).

SUMMARY:
This study is aiming to look into patients' treatment preferences and their socio economic background as well as the exploration of thought processes leading to these preferences. It will integrate, in two exploratory questionnaires, the three most common treatment schema (standard of care, non-operative management, surgery alone) all of which have been demonstrated efficacious.

DETAILED DESCRIPTION:
The primary study objective is to evaluate socioeconomic and demographic factors involved in patients' / physicians treatment preferences. The secondary objective is to assess the tradeoff level between the benefits versus quality of life.

This study will evaluate 192 participants: 14 physicians (group A) and 178 patients (group B).

Participants with operable rectal cancer or health professionals will be screened for eligibility. Subsequently, these participants will be offered to participate in this pilot study and provided a consent form. When a participant has consented to participate, he/she will be provided with a first questionnaire (socio-demographic characteristics, some clinical data and medical baseline information as well as details about their current knowledge about treatments).

An informational brochure will be given after answering the first questionnaire describing different treatment regimens, treatment duration, potential side effects and oncologic outcomes.

A second questionnaire will be provided (evaluating patients treatment preferences and tradeoff).

The consent form, brochure and questionnaires will be available only in an electronic format (Microsoft Form).

ELIGIBILITY:
Inclusion Criteria:

Group A

* New rectal cancer patient
* Operable patients
* Capable adults older than 18 years of age
* Capacity to sign a consent form
* Capacity to answer questionnaires on an online platform Group B
* Treating physician specialists
* Capacity to sign a consent form
* Capacity to answer questionnaires on an online platform

Exclusion Criteria:

Group A:

* Patient unable to sign a consent form
* Patients with metastasis
* Recurrent tumours
* Inability to answer questionnaires on an online platform
* Inability to communicate in french or english

Group B:

* Participant unable to sign a consent form
* Inability to answer questionnaires on an online platform

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will evaluate 192 participants:
  * 14 physicians (group A)
  * 178 patients (group B)
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Socio-economic and demographic characteristics | 1 day
  The primary study objective is to evaluate socioeconomic and demographic factors involved in patients' / physicians treatment preferences. This will be evaluated with the first questionnaire given at the time of the first consultation or when first approached by a research team member.

SECONDARY OUTCOMES:
Tradeoff level | 1 day
  The second objective is to assess the tradeoff level between the benefits versus quality of life. This will be evaluated with the second questionnaire given 2-3 weeks after the first consultation or after answering the first questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Té Vuong, Principal Investigator — Lady Davis Institute - JGH
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pieterse AH, Kunneman M, van den Hout WB, Baas-Thijssen M, Geijsen ED, Ceha HM, Muller KM, van der Linden YM, Marijnen CAM, Stiggelbout AM. Patient explicit consideration of tradeoffs in decision making about rectal cancer treatment: benefits for decision process and quality of life. Acta Oncol. 2019 Jul;58(7):1069-1076. doi: 10.1080/0284186X.2019.1594363. Epub 2019 Apr 11. PMID 30971150
- [Background] Saclarides TJ. Transanal Endoscopic Microsurgery. Clin Colon Rectal Surg. 2015 Sep;28(3):165-75. doi: 10.1055/s-0035-1562889. PMID 26491409
- [Background] Maggiori L, Panis Y. Transanal endoscopic microsurgery (TEM) for T1 rectal cancer. Acta Chir Iugosl. 2012;59(2):87-90. doi: 10.2298/aci1202087m. PMID 23373364
- [Background] Cunningham C. Transanal endoscopic microsurgery. Recent Results Cancer Res. 2014;203:31-8. doi: 10.1007/978-3-319-08060-4_4. PMID 25102997
- [Background] Habr-Gama A, Sabbaga J, Gama-Rodrigues J, Sao Juliao GP, Proscurshim I, Bailao Aguilar P, Nadalin W, Perez RO. Watch and wait approach following extended neoadjuvant chemoradiation for distal rectal cancer: are we getting closer to anal cancer management? Dis Colon Rectum. 2013 Oct;56(10):1109-17. doi: 10.1097/DCR.0b013e3182a25c4e. PMID 24022527
- [Background] Garant A, Magnan S, Devic S, Martin AG, Boutros M, Vasilevsky CA, Ferland S, Bujold A, DesGroseilliers S, Sebajang H, Richard C, Vuong T. Image Guided Adaptive Endorectal Brachytherapy in the Nonoperative Management of Patients With Rectal Cancer. Int J Radiat Oncol Biol Phys. 2019 Dec 1;105(5):1005-1011. doi: 10.1016/j.ijrobp.2019.08.042. Epub 2019 Aug 30. PMID 31476417
- [Background] van der Valk MJM, Marijnen CAM, van Etten B, Dijkstra EA, Hilling DE, Kranenbarg EM, Putter H, Roodvoets AGH, Bahadoer RR, Fokstuen T, Ten Tije AJ, Capdevila J, Hendriks MP, Edhemovic I, Cervantes AMR, de Groot DJA, Nilsson PJ, Glimelius B, van de Velde CJH, Hospers GAP; Collaborative investigators. Compliance and tolerability of short-course radiotherapy followed by preoperative chemotherapy and surgery for high-risk rectal cancer - Results of the international randomized RAPIDO-trial. Radiother Oncol. 2020 Jun;147:75-83. doi: 10.1016/j.radonc.2020.03.011. Epub 2020 Mar 30. PMID 32240909
- [Background] van der Valk MJM, van der Sande ME, Toebes RE, Breukink SO, Broker MEE, Doornebosch PG, Maliko N, Neijenhuis PA, Marinelli AWKS, Peters FP, Peeters KCMJ, Beets GL, Marang-van de Mheen PJ, Hilling DE. Importance of patient reported and clinical outcomes for patients with locally advanced rectal cancer and their treating physicians. Do clinicians know what patients want? Eur J Surg Oncol. 2020 Sep;46(9):1634-1641. doi: 10.1016/j.ejso.2020.04.014. Epub 2020 Apr 15. PMID 32336626
- [Background] Kannan S, Seo J, Riggs KR, Geller G, Boss EF, Berger ZD. Surgeons' Views on Shared Decision-Making. J Patient Cent Res Rev. 2020 Jan 27;7(1):8-18. eCollection 2020 Winter. PMID 32002443
- [Background] Bossema ER, Marijnen CA, Baas-Thijssen MC, van de Velde CJ, Stiggelbout AM. Evaluation of the treatment tradeoff method in rectal cancer patients: is surgery preference related to outcome utilities? Med Decis Making. 2008 Nov-Dec;28(6):888-98. doi: 10.1177/0272989X08317013. Epub 2008 Jun 2. PMID 18519887
- [Background] Smith SK, Trevena L, Simpson JM, Barratt A, Nutbeam D, McCaffery KJ. A decision aid to support informed choices about bowel cancer screening among adults with low education: randomised controlled trial. BMJ. 2010 Oct 26;341:c5370. doi: 10.1136/bmj.c5370. PMID 20978060
- [Background] Ryan M, Farrar S. Using conjoint analysis to elicit preferences for health care. BMJ. 2000 Jun 3;320(7248):1530-3. doi: 10.1136/bmj.320.7248.1530. No abstract available. PMID 10834905
- [Background] Pieterse AH, Berkers F, Baas-Thijssen MC, Marijnen CA, Stiggelbout AM. Adaptive Conjoint Analysis as individual preference assessment tool: feasibility through the internet and reliability of preferences. Patient Educ Couns. 2010 Feb;78(2):224-33. doi: 10.1016/j.pec.2009.05.020. Epub 2009 Jul 5. PMID 19581069
- [Background] Pieterse AH, Stiggelbout AM, Marijnen CA. Methodologic evaluation of adaptive conjoint analysis to assess patient preferences: an application in oncology. Health Expect. 2010 Dec;13(4):392-405. doi: 10.1111/j.1369-7625.2010.00595.x. PMID 20550594
- [Background] ANZGOG and PORTEC Group; Blinman P, Mileshkin L, Khaw P, Goss G, Johnson C, Capp A, Brooks S, Wain G, Kolodziej I, Veillard AS, O'Connell R, Creutzberg CL, Stockler MR. Patients' and clinicians' preferences for adjuvant chemotherapy in endometrial cancer: an ANZGOG substudy of the PORTEC-3 intergroup randomised trial. Br J Cancer. 2016 Nov 8;115(10):1179-1185. doi: 10.1038/bjc.2016.323. Epub 2016 Oct 20. PMID 27764842
- [Background] Lee L, Trepanier M, Renaud J, Liberman S, Charlebois P, Stein B, Fried GM, Fiore J Jr, Feldman LS. Patients' preferences for sphincter preservation versus abdominoperineal resection for low rectal cancer. Surgery. 2021 Mar;169(3):623-628. doi: 10.1016/j.surg.2020.07.020. Epub 2020 Aug 24. PMID 32854970
- [Background] Couwenberg AM, Intven MPW, Burbach JPM, Emaus MJ, van Grevenstein WMU, Verkooijen HM. Utility Scores and Preferences for Surgical and Organ-Sparing Approaches for Treatment of Intermediate and High-Risk Rectal Cancer. Dis Colon Rectum. 2018 Aug;61(8):911-919. doi: 10.1097/DCR.0000000000001029. PMID 29697477
- [Background] Stiggelbout AM, Pieterse AH, De Haes JC. Shared decision making: Concepts, evidence, and practice. Patient Educ Couns. 2015 Oct;98(10):1172-9. doi: 10.1016/j.pec.2015.06.022. Epub 2015 Jul 15. PMID 26215573
- [Background] Kunneman M, Marijnen CA, Baas-Thijssen MC, van der Linden YM, Rozema T, Muller K, Geijsen ED, Stiggelbout AM, Pieterse AH. Considering patient values and treatment preferences enhances patient involvement in rectal cancer treatment decision making. Radiother Oncol. 2015 Nov;117(2):338-42. doi: 10.1016/j.radonc.2015.09.005. Epub 2015 Sep 11. PMID 26372343
- [Background] Snijders HS, Kunneman M, Bonsing BA, de Vries AC, Tollenaar RA, Pieterse AH, Stiggelbout AM. Preoperative risk information and patient involvement in surgical treatment for rectal and sigmoid cancer. Colorectal Dis. 2014 Feb;16(2):O43-9. doi: 10.1111/codi.12481. PMID 24188458
- [Background] Kunneman M, Engelhardt EG, Ten Hove FL, Marijnen CA, Portielje JE, Smets EM, de Haes HJ, Stiggelbout AM, Pieterse AH. Deciding about (neo-)adjuvant rectal and breast cancer treatment: Missed opportunities for shared decision making. Acta Oncol. 2016;55(2):134-9. doi: 10.3109/0284186X.2015.1068447. Epub 2015 Aug 3. PMID 26237738
- [Background] Pieterse AH, Henselmans I, de Haes HC, Koning CC, Geijsen ED, Smets EM. Shared decision making: prostate cancer patients' appraisal of treatment alternatives and oncologists' eliciting and responding behavior, an explorative study. Patient Educ Couns. 2011 Dec;85(3):e251-9. doi: 10.1016/j.pec.2011.05.012. Epub 2011 Jun 11. PMID 21658883
- [Background] Pieterse AH, Kunneman M, Engelhardt EG, Brouwer NJ, Kroep JR, Marijnen CAM, Stiggelbout AM, Smets EMA. Oncologist, patient, and companion questions during pretreatment consultations about adjuvant cancer treatment: a shared decision-making perspective. Psychooncology. 2017 Jul;26(7):943-950. doi: 10.1002/pon.4241. Epub 2016 Sep 15. PMID 27502561
- [Background] Pieterse AH, de Vries M, Kunneman M, Stiggelbout AM, Feldman-Stewart D. Theory-informed design of values clarification methods: a cognitive psychological perspective on patient health-related decision making. Soc Sci Med. 2013 Jan;77:156-63. doi: 10.1016/j.socscimed.2012.11.020. Epub 2012 Nov 27. PMID 23219164
- [Background] Fagerlin A, Pignone M, Abhyankar P, Col N, Feldman-Stewart D, Gavaruzzi T, Kryworuchko J, Levin CA, Pieterse AH, Reyna V, Stiggelbout A, Scherer LD, Wills C, Witteman HO. Clarifying values: an updated review. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S8. doi: 10.1186/1472-6947-13-S2-S8. Epub 2013 Nov 29. PMID 24625261
- [Background] Munro S, Stacey D, Lewis KB, Bansback N. Choosing treatment and screening options congruent with values: Do decision aids help? Sub-analysis of a systematic review. Patient Educ Couns. 2016 Apr;99(4):491-500. doi: 10.1016/j.pec.2015.10.026. Epub 2015 Nov 2. PMID 26549169
- [Background] Papaccio F, Rosello S, Huerta M, Gambardella V, Tarazona N, Fleitas T, Roda D, Cervantes A. Neoadjuvant Chemotherapy in Locally Advanced Rectal Cancer. Cancers (Basel). 2020 Dec 3;12(12):3611. doi: 10.3390/cancers12123611. PMID 33287114
- [Background] Nilsson PJ, van Etten B, Hospers GA, Pahlman L, van de Velde CJ, Beets-Tan RG, Blomqvist L, Beukema JC, Kapiteijn E, Marijnen CA, Nagtegaal ID, Wiggers T, Glimelius B. Short-course radiotherapy followed by neo-adjuvant chemotherapy in locally advanced rectal cancer--the RAPIDO trial. BMC Cancer. 2013 Jun 7;13:279. doi: 10.1186/1471-2407-13-279. PMID 23742033
- [Background] Bahadoer RR, Dijkstra EA, van Etten B, Marijnen CAM, Putter H, Kranenbarg EM, Roodvoets AGH, Nagtegaal ID, Beets-Tan RGH, Blomqvist LK, Fokstuen T, Ten Tije AJ, Capdevila J, Hendriks MP, Edhemovic I, Cervantes A, Nilsson PJ, Glimelius B, van de Velde CJH, Hospers GAP; RAPIDO collaborative investigators. Short-course radiotherapy followed by chemotherapy before total mesorectal excision (TME) versus preoperative chemoradiotherapy, TME, and optional adjuvant chemotherapy in locally advanced rectal cancer (RAPIDO): a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):29-42. doi: 10.1016/S1470-2045(20)30555-6. Epub 2020 Dec 7. PMID 33301740
- [Background] Smith JJ, Chow OS, Gollub MJ, Nash GM, Temple LK, Weiser MR, Guillem JG, Paty PB, Avila K, Garcia-Aguilar J; Rectal Cancer Consortium. Organ Preservation in Rectal Adenocarcinoma: a phase II randomized controlled trial evaluating 3-year disease-free survival in patients with locally advanced rectal cancer treated with chemoradiation plus induction or consolidation chemotherapy, and total mesorectal excision or nonoperative management. BMC Cancer. 2015 Oct 23;15:767. doi: 10.1186/s12885-015-1632-z. PMID 26497495